CLINICAL TRIAL: NCT02151825
Title: Pilot Study on the Influence of a Synbiotic Formulation (ProSynbiotic) on Gut Microbiota Composition, Adiposity and Selected Markers of Cardiometabolic Health in Overweight or Moderately Obese Individuals
Brief Title: Effect of a Synbiotic on the Gut Microbiota and Adiposity-related Markers in Healthy Overweight Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas State University, San Marcos (Other)
Collaborators: Standard Process Inc. (Industry)
Responsible Party: Principal Investigator, Vatsala Maitin, Assistant Professor, Texas State University, San Marcos
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2011F7611; 110021 (Other: Texas State University)
Record Dates: First submitted 2014-05-28; First posted 2014-05-30 (Estimated); Last update posted 2014-05-30 (Estimated); Status verified 2014-05

CONDITIONS: Gut Microbiota; Adiposity
Keywords: Gut microbiota; Probiotics; Prebiotics; Synbiotic; Bifidobacterium lactis BB-12; Lactobacillus acidophilus LA-5; Lactobacillus casei 431; Inulin; GOS; Body Weight; Overweight; Adiposity; Obesity; ANGPTL4
MeSH Terms: conditions — Obesity; Body Weight; Overweight | interventions — Synbiotics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Synbiotic (Experimental): 3 capsules per day containing 4 billion CFU of Bifidobacterium lactis BB-12, Lactobacillus acidophilus LA-5, Lactobacillus casei 431 and Saccharomyces boulardii in combination with prebiotics Inulin (1 g) and Galactooligosaccharides (100 mg)
  Interventions: Dietary Supplement: Synbiotic
- Placebo (Placebo Comparator): 3 capsules of Maltodextrin per day
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Synbiotic — 3 capsules per day containing 4 billion CFU of Bifidobacterium lactis BB-12, Lactobacillus acidophilus LA-5, Lactobacillus casei 431 and Saccharomyces boulardii in combination with prebiotics Inulin (1 g) and Galactooligosaccharides (100 mg)
  Other Names: Prosynbiotic
  Arms: Synbiotic
Other: Placebo — 3 capsules of Maltodextrin per day
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the effects of a synbiotic (ProSynbiotic) on the gut microbiota composition, body composition and adiposity-related genes and metabolic markers in healthy overweight adult subjects.

DETAILED DESCRIPTION:
This is a parallel, double-blind, randomized, placebo controlled trial to determine the effects of a synbiotic formulation (ProSynbiotic) containing 4 billion CFU of a probiotic blend of Bifidobacterium lactis BB-12, Lactobacillus acidophilus LA-5, Lactobacillus casei 431 and Saccharomyces boulardii, along with 1 g of the prebiotic inulin and 100 mg of galactooligosaccharide (GOS) on the gut microbiota composition, body composition, expression of genes mediating dietary energy harvest and adiposity, and on adiposity-related metabolic markers in healthy free-living overweight or moderately obese subjects. The duration of the study is 18 weeks, including a 2-week run-in period before randomization of subjects into the synbiotic or placebo group, a 12-week intervention period, and a 4-week follow-up after the end of the intervention. During the intervention period, subjects will be instructed to take 3 capsules of either synbiotic or placebo per day and maintain their habitual diet and physical activity. They will also be asked to document any unusual symptoms or side effects as well as keep a bowel diary. Diet and physical activity will be monitored via 24-h dietary recalls and the global physical activity questionnaire respectively. Changes in the gut microbiota composition will be determined by measuring bacterial population levels in stool sampled collected at baseline, 6 weeks, 12 weeks and the follow up time point. Body composition will be measured using the BOD POD at baseline, 6 weeks, and 12 weeks. Gene expression levels will be assessed at baseline and 12 weeks in colonocytes (isolated from stool samples) and PBMCs (isolated from blood samples) by qPCR. Metabolic markers will be measured at baseline and 12-weeks in plasma or serum using the respective biochemical- or immuno-assays.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-64
* BMI of 25-34.9 and/or a waist circumference >35 inches for women and >40 inches for men
* Generally healthy except for overweight or moderately obese
* A signed consent form
* Passed a screening questionnaire and willingness to comply with study procedures
* Lipid levels, fasting glucose, liver function and complete blood counts within the normal reference ranges as measured in a screening blood sample

Exclusion Criteria:

* Persons on a weight-loss regimen
* Antibiotic use (< 3 months before the study)
* Regular probiotic, prebiotic or synbiotic use (< 1 month before the study)
* Regular use of anti-inflammatory drugs, weight-loss medications or supplements (< 1 month prior to the study)
* Personal history of cardiovascular disease, hypertension, cancer, type 1 or type 2 diabetes and inflammatory gastrointestinal disorders such as Crohn's disease or colitis
* Smoking
* Consumption of >2 units of alcohol per day
* Pregnancy or lactation
* Irregular periods, menopause or hormone replacement therapy
* Over 300 minutes of exercise per week

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2011-09; Primary Completion 2012-09 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Changes to the gut microbiota | 0-weeks (Baseline), 6-weeks (midpoint of intervention), 12-weeks (end of intervention) and 16-weeks (4-weeks after end of intervention)
  The primary objective of this study is to determine the effect of a synbiotic formulation called ProSynbiotic (administered at 3 capsules/day) containing 4 billion CFU of a probiotic blend of Bifidobacterium lactis BB-12, Lactobacillus acidophilus LA-5, Lactobacillus casei 431 and Saccharomyces boulardii, along with 1 g of the prebiotic inulin and 100 mg of galactooligosaccharide (GOS) on the gut microbiota of healthy overweight adult subjects when compared to a placebo of maltodextrin. Changes in the gut microbiota will be determined by measuring specific bacterial population levels in the subjects' fecal samples, using 16S rRNA targeted oligonucleotide probes and fluorescence in situ hybridisation.

SECONDARY OUTCOMES:
Body composition | Baseline, 6-weeks and 12-weeks.
  The effect of Prosynbiotic on the subjects' body composition will be evaluated by BOD POD assessment carried out at baseline, 6-weeks and 12-weeks.
Expression of genes mediating dietary energy harvest and adiposity | Baseline and 12-weeks
  This will be achieved by measuring the gene expression levels of ANGPTL4, PPAR-γ and GPR41/43 in colonocytes isolated from stool and that of ANGPTL4, PPAR-γ, NF-kB, IL-6 and TNF-α in PBMCs isolated from blood collected from the subjects at baseline and 12-weeks.
Adiposity-related metabolic markers | Baseline and 12-weeks
  This will be achieved by measuring TNF-α, adiponectin, total cholesterol, LDL-C, HDL-C, triglycerides and glucose levels in fasting blood samples collected from the study subjects at baseline and 12-weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Vatsala Maitin, PhD, Principal Investigator — Texas State University
Locations (1):
- Texas State University, San Marcos, Texas, United States